CLINICAL TRIAL: NCT03296943
Title: A Novel Approach of Substitution Therapy With Inhalation of Essential Oil for the Reduction of Inhalants Craving: A Double-blinded Randomized Controlled Trial
Brief Title: Efficacy of Inhalation of Essential Oil on the Reduction of Inhalants Craving
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Rasmon Kalayasiri, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Graduate School Grant 2553
Record Dates: First submitted 2017-09-24; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Inhalants Craving
MeSH Terms: interventions — Oils, Volatile; Perfume

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The containers for essential oil and perfume are identical dark-glass tubes with a roll-on-cap on top and double-covered with a plain cap on each tube.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essential oil (Experimental): Essential oil is prepared from the product of Thailada with manufacture standard ID 1087/2548 by Thailand Ministry of Industry. Essential oil is extracted by a cold compressed method from the lavandula angustifolia (lavender) grown in Australia.
  Interventions: Combination Product: Essential oil; Behavioral: Cue-induced inhalants craving
- Perfume (Sham Comparator): Perfume is the synthetic perfume of lavender flavor without essential oil.
  Interventions: Combination Product: Perfume; Behavioral: Cue-induced inhalants craving

INTERVENTIONS:
Combination Product: Essential oil — To inhale the essential oil in an air-conditioned room, the container was flipped over to soak the roll-on cap that was then rolled-on circularly at the right mid-palm of the subject at 2 centimeter in diameter for 5 cycles.
  Arms: Essential oil
Combination Product: Perfume — To inhale the perfume in an air-conditioned room, the container was flipped over to soak the roll-on cap that was then rolled-on circularly at the right mid-palm of the subject at 2 centimeter in diameter for 5 cycles.
  Arms: Perfume
Behavioral: Cue-induced inhalants craving — Exposing individuals with a set of 12 pictures for one-minute (e.g., 5 second display per picture) every five minutes for three sets in total followed by another three sets of neutral/relaxing pictures of nature.

SUMMARY:
Inhalants, which are neurotoxic central nervous system (CNS) suppressants, are frequently abused by young adults. Unlike other CNS depressants, including alcohol and opiates, no treatment is currently approved for inhalants dependence. In this report, a novel approach of substitution treatment for inhalants addiction was explored in a double-blinded, randomized, controlled crossover design to examine the effects of inhalation of essential oil (EO) and perfume (PF) on the reduction of cue-induced craving for inhalants in a cohort of thirty-four Thai males with inhalants dependence. The craving response was measured by the modified version of Penn Alcohol Craving Score for Inhalants (PACS-inhalants)

ELIGIBILITY:
Inclusion Criteria:

* Participants with ability to smell if they could correctly identify 3 out of 5 odors, namely fish sauce, lemon, onion, basil, and jasmine.
* Individuals with inducible picture-cues inhalant craving based on a 50% increase in craving score from baseline.

Exclusion Criteria:

* Individuals with a history of major psychiatric disorders, including psychotic and mood disorders
* Individuals with illicit substance dependence other than inhalants
* Individuals with allergic reactions to essential oil or perfume.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2010-11-30 (Actual)

PRIMARY OUTCOMES:
Inhalants craving - PACS | Daily for 3 days
  Inhalants craving was measured by the Penn Alcohol Craving Scale for Inhalants (PACS-inhalants)
Inhalants craving - VAS | Daily for 3 days
  Inhalants craving was measured by the Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Rasmon Kalayasiri, M.D., Principal Investigator — Chulalongkorn University Faculty of Medicine
Locations (1):
- Princess Mother National Institute on Drug Abuse Treatment, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No